CLINICAL TRIAL: NCT05273073
Title: Roles of Probiotics on Gut Microbiata Composition and Metabolic Outcomes in Women With a Recent History of Gestational Diabetes Mellitus: A Randomised Control Trial
Brief Title: Effects of Probiotics on Gut Microbiota Composition and Metabolic Outcomes in Post- Gestational Diabetes Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: B-Crobes Laboratory (M) Sdn Bhd (Unknown); Ministry of Higher Education, Malaysia (Other)
Responsible Party: Principal Investigator, PROF DR RAJA AFFENDI RAJA ALI, Consultant Physician & Gastroenterologist, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UKM PPI/111/8/JEP-2018-022; AP-2017-008/2 (Other Grant/Funding Number: Ministry of Higher Education, Malaysia)
Record Dates: First submitted 2022-02-18; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; probiotics; gut microbiota; glycemic control
MeSH Terms: conditions — Diabetes, Gestational | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This was a 12-week randomized, double-blind, placebo-controlled, parallel-group clinical trial in post-gestational diabetes women. Participants were randomly received either placebo or 30 billion colony forming units of probiotics (HEXBIO® Microbial Cell Preparation, MCP® BCMC® Strains) consist of six viable microorganisms of Lactobacillus and Bifidobacteria strains, twice daily for 12-week.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Active Comparator): 83 participants received probiotics for 12-week
  Interventions: Dietary Supplement: Probiotics
- Placebo group (Placebo Comparator): 83 participants received placebo for 12-week
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Each sachet consists of 30 billion colony-forming units (CFU) of six viable probiotic strains (Lactobacillus acidophilus BCMC® 12130 (107 mg), Lactobacillus casei subsp. BCMC® 12313 (107 mg), Lactobacillus lactis BCMC® 12451 (107 mg), Bifidobacterium bifidum BCMC® 02290 (107 mg), Bifidobacterium infantis BCMC® 02129 (107 mg), and Bifidobacterium longum BCMC® 02120 (107 mg).
  Other Names: HEXBIO® Microbial Cell Preparation (MCP)
  Arms: Probiotics group
Dietary Supplement: Placebo — Placebo samples were identical to the probiotics in term of taste and texture without live microbial cells.
  Arms: Placebo group

SUMMARY:
Risk of developing diabetes at a younger age among women with a previous history of gestational diabetes mellitus (post-GDM) has increased by 10-fold compared to the healthy women. However, consistent long-term lifestyle modifications by diet restriction and exercise are challenging. Interestingly, probiotics were found to balance gut bacteria and improve host metabolism. Thus, the aim of this study is to determine the beneficial roles of probiotics supplementation in post-GDM women.

DETAILED DESCRIPTION:
Recent evidence highlighted disturbances in gut microbial compositions were associated with impairment of glucose and inflammation metabolism in women with GDM. Probiotics were hypothesized will modulate gut microbial compositions and maintain glucose and inflammation in the post-GDM women. This study aims to elucidate the roles of probiotic supplementation on metabolic and inflammatory outcomes in women with a previous history of gestational diabetes mellitus.

This is a 12-week randomized, double-blind, placebo-controlled, parallel-group clinical trial involving participants who had attended postnatal follow-up at Universiti Kebangsaan Malaysia Medical Centre (UKMMC) with a recent history of GDM and had either postpartum glucose intolerance or overweight (body mass index (BMI) ≥23 kg/m2), or obese (BMI ≥27.5 kg/m2) during eligibility assessment.

A total of 166 post-GDM participants with either postpartum glucose intolerance or overweight/obese were randomly assigned to probiotics (n = 83) and placebo (n= 83) groups. Eligible participants were given probiotics supplementation consisting of 30 billion colony forming units (CFU) of six viable microorganisms from Lactobacillus and Bifidobacteria strains, twice daily for 12-week.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years.
* Attended postnatal follow-up at Universiti Kebangsaan Medical Center (four to eight weeks postpartum).
* Have a recent history of gestational diabetes mellitus.
* Willing to participate in the study.
* Had either postpartum glucose intolerance, overweight (BMI ≥23 kg/m2), or obese (BMI ≥27.5 kg/m2) during eligibility assessment.

Exclusion Criteria:

* Postpartum fasting blood glucose (FBG) level >8.0 mmol/L, two-hour postprandial (2HPP) glucose level >12 mmol/L.
* Symptomatic of hyperglycemia and started on hypoglycemic agent.
* Have underlying medical illnesses and required regular medications (i.e., pre- pregnancy diabetes, hypertension, congestive heart failure, renal failure, liver cirrhosis, gastrointestinal diseases, autoimmune diseases, and cancer) before and during intervention.
* Had taken antibiotics / regularly consumed food or supplements rich in prebiotics/probiotics/symbiotics less than 12-week before recruitment or during intervention.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with a recent history of gestational diabetes mellitus
Enrollment: 166 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Mean difference of fasting blood glucose (FBG) | 12-week
  Fasting blood glucose (FBG) levels were measured at the baseline and at the end of trial (post-12 weeks intervention). The mean difference of FBG was obtained by comparing the FBG levels at the end of trial with FBG levels at baseline. The mean difference of FBG levels were assessed within each intervention group and between the two intervention groups.
Mean difference of HbA1c | 12-week
  HbA1c levels at the baseline and at the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.
Mean difference of fasting serum insulin (FSI) | 12-week
  FSI levels at the baseline and at the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.
Mean difference of glucagon-like peptide -1 (GLP-1 active) | 12-week
  GLP-1 active levels at the baseline and the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.
Mean difference of homeostasis model assessment of insulin resistance (HOMA-IR) | 12-week
  HOMA-IR levels at the baseline and at the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.

SECONDARY OUTCOMES:
Mean difference of body mass index (BMI) | 12-week
  The detail for height was obtained from the antenatal record. The weight of participants at the baseline and the end of the trial (post-12 weeks intervention) was measured. BMI was calculated by dividing body weight (kg) with the square of the height (m2). BMI was compared within each intervention group and between the two intervention groups
Mean difference of waist circumference | 12-week
  Waist circumference at the baseline and the end of the trial (post-12 weeks intervention) was measured and compared within each intervention group and between the two intervention groups
Mean difference of blood pressure | 12-week
  Systolic and diastolic blood pressure at the baseline and the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups
Mean difference of total cholesterol and triglycerides | 12-week
  Total cholesterol and triglycerides levels at the baseline and the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.
Mean difference of high sensitivity-C reactive protein (hs-CRP) | 12-week
  hs-CRP at the baseline and the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.
Mean difference of other inflammatory markers (interleukin-1β, IL-6, and IL-8) | 12-week
  IL-1β, IL-6, and IL-8 levels at the baseline and the end of the trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.
Changes in gut microbial profiles (i.e., gut microbial composition, alpha diversity, beta diversity, and functional analysis) | 12-week
  Gut microbial composition, alpha diversity, beta diversity, and functional analysis at the baseline and at the end of trial (post-12 weeks intervention) were measured and compared within each intervention group and between the two intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr. Raja Affendi Raja Ali, Principal Investigator — Gastroenterology Unit, Faculty of Medicine, Universiti Kebangsaan Malaysia, Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No